CLINICAL TRIAL: NCT05695482
Title: Progressive Resistance Training Compared to Neuromuscular Exercises on Knee Kinematics in Two Functional Tests. Α Single-blinded Randomised Controlled Trial Protocol.
Brief Title: Progressive Resistance Training Compared to Neuromuscular Exercises on Knee Kinematics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Savvas Spanos, Director of Human Performance and Rehabilitation Laboratory of the Physiotherapy Department, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2023-01-10; First posted 2023-01-25 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Dynamic Knee Valgus; Injury Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular exercise training (NMT) (Experimental): The 6-week exercise intervention consists of group sessions of Neuromuscular training supervised by a researcher 3 times per week. Participants will be familiarized with the exercises on a separate day prior to testing.
  Each session consists of a 5-minute submaximal warm-up followed by 25 minutes of NM training with closed kinetic chain exercises.
  Every 2 weeks, there will be a progression that will be achieved by increasing the level of difficulty of each the exercise. We will take into consideration when an exercise is performed with appropriate sensorimotor control, quality of the performance, minimal exertion and control of the movement. Participants will be given special equipment including a step measuring 20 cm in height, an uneven surface, a slider and an elastic tubing medium load (green) from Thera BandTM, (Akron, Ohio, USA).
  Interventions: Other: Neuromuscular training exercises
- Progressive Resistance Training (PRT) (Experimental): The 6-week exercise intervention consists of group sessions of progressive resistance training supervised by a researcher 3 times per week. Participants will be familiarized with the exercises on a separate day prior to testing.
  Each session consists of a 5-minute submaximal warm-up followed by 20 minutes of PRT with an open kinetic chain (no weight-bearing exercises) targeting the abductors' muscles of the hip joint. The exercise intensity will be monitored by the researcher, as determined by the patient's ability to complete three sets of 8-12 repetitions for a given exercise and a Borg Rating of Perceived Exertion (RPE) of 6-8.
  Every 2 weeks, there will be a progression achieved by changing the resistance in line with guidelines provided by the American College of Sports Medicine with an elastic tubing heavy load (grey) from Thera BandTM, (Akron, Ohio, USA)
  Interventions: Other: Hip abductors muscular strength exercises

INTERVENTIONS:
Other: Neuromuscular training exercises — The 6-week exercise intervention consists of 25-minute group sessions of Neuromuscular training supervised by a researcher.
  Arms: Neuromuscular exercise training (NMT)
Other: Hip abductors muscular strength exercises — The 6-week exercise intervention consists of of 20-minute group sessions of progressive resistance training, supervised by a researcher.
  Arms: Progressive Resistance Training (PRT)

SUMMARY:
The primary aim of this randomized controlled trial is to investigate the effectiveness of 6 weeks of progressive resistance training (PRT) compared to neuromuscular training (NMT) on functional performance in healthy female participants as measured by the Single-Leg Landing (SLL) and Single-Leg Squat (SLS) tests.

The secondary aims are to investigate the,

* change in abduction hip muscle strength, which will be measured with a Biodex System 3 Isokinetic Dynamometer. Outcomes will be measured at baseline and after 6 weeks of intervention.
* adherence to the 6-week initial intervention (High adherence is defined as ≥ 80% attendance to the supervised interventions.)

DETAILED DESCRIPTION:
Participants will be randomized into two groups: PRT or NMT. Outcomes will be measured at baseline and after 6 weeks of intervention.

All sessions will be conducted in group sessions, with one researcher supervising the exercises. Patients receive education as well as supervised exercise from trained physiotherapists. Each session will last approximately 25-30 minutes. The duration of the program will be 6 weeks, with 3 sessions every week (total: 18 training sessions).

The NMT intervention sessions consist of a 5-minute submaximal warm-up followed by 25 minutes of NMT training with exercises focused on functional stability, proprioception, strength, stability, agility, postural function, and postural orientation. The training sessions will consist of two parts: warming up and the circuit program. The circuit program will consist of 8 exercises. Each exercise will be performed for 2 sets of 10 repetitions, with a rest of 30 sec corresponding to every set, between each set and exercises. The exercises will be focused on one knee, which will then be evaluated. Three levels of difficulty will be given for each exercise to allow for progression. Every 2 weeks, there will be a progression that will be achieved by changing the exercise and gradually making it harder, or/and changing the support surface.

In the PRT intervention, the sessions will consist of a 5-minute submaximal warm-up followed by 20 minutes of PRT with exercises targeting the abductor muscles of the hip joint. The circuit program will consist of three exercises. Each exercise will be performed in sets of three, then increased to four sets of ten repetitions, with a 30-second rest between each set and exercise.

The exercise intensity will be monitored by the researcher, as determined by the patient's ability to complete three sets of 8-12 repetitions for a given exercise and a Borg Rating of Perceived Exertion (RPE) of 6-10. The progression will be in line with guidelines provided by the American College of Sports Medicine.

Adherence to the program for both groups will be assessed by the total number of training sessions performed in 6 weeks (total = 18 training sessions).

ELIGIBILITY:
Inclusion Criteria:

* female gender
* older than 18 and younger than 35 years of age
* physically able to perform physical activities and exercise
* participants should know the greek language in order to understand the instructions and be able to read the consent form

Exclusion Criteria:

* undergoing treatment for lower extremity injury
* currently experiencing an average overall pain severity ≥3 out of 10 on an 11-point numerical rating scale in the past week
* history of knee pain in the proceeding twelve months, history of lower limb surgery, known rheumatologic, neurological or cardiovascular disorders with raised blood pressure

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Changes in knee kinematics measured during a Single-Leg Squat functional test | Measured at baseline and Week 6.
  Dynamic Knee Valgus (recorded in degrees) will be assessed during a Single-Leg Squat test. Changes during the test will be analyzed with the Kinovea program.
Changes in knee kinematics measured during a Single-Leg Landing functional test | Measured at baseline and Week 6.
  Dynamic Knee Valgus (recorded in degrees) will be assessed during a Single-Leg Landing test. Changes during the test will be analyzed with the Kinovea program.

SECONDARY OUTCOMES:
Change in abduction hip muscle power | Measured at baseline and Week 6.
  Change in abduction hip muscle power (measured in Newtons) will be measured with a Biodex System 3 isokinetic dynamometer.
Adherence to the 6-week initial intervention | Measured at Week 6.
  High adherence is defined as ≥ 80% attendance to the supervised interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Thessaly, Lamia, Central Greece, Greece

REFERENCES:
- [Background] Kraemer WJ, Adams K, Cafarelli E, Dudley GA, Dooly C, Feigenbaum MS, Fleck SJ, Franklin B, Fry AC, Hoffman JR, Newton RU, Potteiger J, Stone MH, Ratamess NA, Triplett-McBride T; American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2002 Feb;34(2):364-80. doi: 10.1097/00005768-200202000-00027. PMID 11828249
- [Background] Ageberg E, Roos EM. Neuromuscular exercise as treatment of degenerative knee disease. Exerc Sport Sci Rev. 2015 Jan;43(1):14-22. doi: 10.1249/JES.0000000000000030. PMID 25390299
- [Background] Day ML, McGuigan MR, Brice G, Foster C. Monitoring exercise intensity during resistance training using the session RPE scale. J Strength Cond Res. 2004 May;18(2):353-8. doi: 10.1519/R-13113.1. PMID 15142026
- [Background] Peixoto Leao Almeida G, Oliveira Monteiro I, Larissa Azevedo Tavares M, Lourinho Sales Porto P, Rocha Albano T, Pasqual Marques A. Hip abductor versus adductor strengthening for clinical outcomes in knee symptomatic osteoarthritis: A randomized controlled trial. Musculoskelet Sci Pract. 2022 Oct;61:102575. doi: 10.1016/j.msksp.2022.102575. Epub 2022 May 13. PMID 35780637
- [Background] Horsak B, Artner D, Baca A, Pobatschnig B, Greber-Platzer S, Nehrer S, Wondrasch B. The effects of a strength and neuromuscular exercise programme for the lower extremity on knee load, pain and function in obese children and adolescents: study protocol for a randomised controlled trial. Trials. 2015 Dec 23;16:586. doi: 10.1186/s13063-015-1091-5. PMID 26700568
- [Background] Bennell KL, Kyriakides M, Metcalf B, Egerton T, Wrigley TV, Hodges PW, Hunt MA, Roos EM, Forbes A, Ageberg E, Hinman RS. Neuromuscular versus quadriceps strengthening exercise in patients with medial knee osteoarthritis and varus malalignment: a randomized controlled trial. Arthritis Rheumatol. 2014 Apr;66(4):950-9. doi: 10.1002/art.38317. PMID 24757146
- [Background] Clausen B, Holsgaard-Larsen A, Roos EM. An 8-Week Neuromuscular Exercise Program for Patients With Mild to Moderate Knee Osteoarthritis: A Case Series Drawn From a Registered Clinical Trial. J Athl Train. 2017 Jun 2;52(6):592-605. doi: 10.4085/1062-6050-52.5.06. PMID 28653869
- [Background] Stefanouli V, Kapreli E, Anastasiadi E, Nakastsis A, Strimpakos N. Validity and reliability of the Greek version of modified Baecke questionnaire. Public Health. 2022 Feb;203:58-64. doi: 10.1016/j.puhe.2021.11.017. Epub 2022 Jan 13. PMID 35032916
- [Background] Palmer K, Hebron C, Williams JM. A randomised trial into the effect of an isolated hip abductor strengthening programme and a functional motor control programme on knee kinematics and hip muscle strength. BMC Musculoskelet Disord. 2015 May 3;16:105. doi: 10.1186/s12891-015-0563-9. PMID 25935843